CLINICAL TRIAL: NCT01921790
Title: An Open-Label, Uncontrolled, Single Centered Phase Ⅱ Study of Avastin Combined With Gemcitabine, Oxaliplatin, Pegaspargase and Dexamethasone (Avastin+ GemAOD) As First-Line Treatment in Patients With Untreated NK/T Cell Lymphoma
Brief Title: Avastin+ GemAOD As First-Line Treatment in NK/T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Hoffmann-La Roche (Industry); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Li Zhiming, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2013-017-01
Record Dates: First submitted 2013-08-03; First posted 2013-08-13 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Extranodal NK/T-cell Lymphoma, Nasal Type
Keywords: Avastin+ GemAOD; first line chemotherapy; NK/T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Bevacizumab; Gemcitabine; Oxaliplatin; pegaspargase; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avastin+ GemAOD (Experimental): Avastin+ GemAOD means Avastin Combined With Gemcitabine, Oxaliplatin, Pegaspargase and Dexamethasone
  Interventions: Biological: Avastin; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Pegaspargase; Drug: Dexamethasone

INTERVENTIONS:
Biological: Avastin — Avastin 7.5mg/Kg, intravenous drip D1
Drug: Gemcitabine — Gemcitabine 1g/m2 intravenous drip D1,D8
Drug: Oxaliplatin — Oxaliplatin 130mg/m2 intravenous drip D1
Drug: Pegaspargase — Pegaspargase 2500U/m2 intramuscular injection (IM) D1
Drug: Dexamethasone — Dexamethasone 20mg/d intravenous drip D1, po D2-3

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of avastin combined with gemcitabine, oxaliplatin, pegaspargase and dexamethasone(Avastin+ GemAOD) as first-line treatment in patients with untreated natural killer(NK)/T cell lymphoma

DETAILED DESCRIPTION:
Recent study showed that vascular endothelial growth factor (VEGF) was associated with a poorer outcome in patients with Non-Hodgkin's Lymphoma,and Avastin impacted on tumor endothelial cells to make standard chemotherapy work better for T cell lymphoma. Many researches on Gemcitabine combined with Oxaliplatin for treatments of recurrent and refractory Non-Hodgkin's lymphoma showed patients could benefit from the combination treatment . Pegaspargase plays an important role for treatment of NK/T cell lymphoma. Dexamethasone is used in combination with other agents for the treatment of lymphomas which may be implicated in the development or growth of some cancers.So we explored to evaluate the efficacy and safety of Avastin combined with gemcitabine, oxaliplatin, pegaspargase and dexamethasone(Avastin+ GemAOD) as first-line treatment in patients with untreated NK/T cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of NK/T Cell Lymphoma;
* Age:18-80 years;
* Eastern Cooperative Oncology Group (ECOG) status 0-3, Estimated survival time > 3 months;
* Normal haematological, liver and renal function (WBC count≥4×109/L, Hemoglobin≥100g/L, platelet count≥100×109/L, bilirubin<1.5×ULN, Alanine transaminase (ALT) or Aspartate Aminotransferase (AST)<2.5×ULN, serum creatinine<1.5×ULN), normal coagulation function and cardiac function;
* Appreciable and measurable lesions ;
* No history of other malignancies;
* No previous treatments including chemotherapy, radiotherapy, targeted therapy or stem cell transplantation;
* No other serious diseases which conflict with the treatment in the present trial;
* No concurrent treatments that conflict with the treatments in the present trial(including steroid drugs);
* Voluntary participation and signed the informed consent.

Exclusion Criteria:

* The patients had the conditions below: clinically significant ventricular tachycardia (VT), atrial fibrillation (AF), heart block, myocardial infarction (MI), congestive heart failure (CHF), symptomatic coronary artery heart disease requiring medication;
* The patients suffered from organ transplant
* The patients participated in other clinical trials within the 30 days before enrollment or who are participating in other clinical studies;
* The patients with active bleeding or new thrombotic disease, who are taking anticoagulant drugs or with a history of bleeding tendencies;
* The patients suffered before surgery less than four weeks, or after less than six weeks;
* The patients with major vascular invasion;
* The patients with abnormal liver function (total bilirubin> 1.5 times the normal value, ALT / AST> 2.5 times normal), abnormal renal function (serum creatinine> 1.5 times normal), blood abnormalities (absolute neutrophil count <1.5 × 109 / L, platelets <80 × 109 / L, hemoglobin <90g /L) ;
* The patients with moderate to severe proteinuria;
* Severe hypertension,BP≥160/100mmHg;
* The patients with mentally ill / unable to obtain informed consent;
* The patients with drug addiction, alcohol abuse which affects the long-term evaluation of test results;
* The patients in pregnancy, lactation and women of childbearing age who do not want to take contraceptive measures subjects;
* Clinical and laboratory support brain metastases;
* The patients with a history of allergy to test drug;
* The patients not suitable to participate in the investigator judged by researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate(ORR) | every 6 weeks,up to completion of treatment(approximately 6 months)
  21 days(3 weeks) for one cycle,Efficacy was evaluated every two cycles

SECONDARY OUTCOMES:
Progress Free Survival(PFS) | up to end of follow-up-phase (approximately 5 years)
Overall Survival(OS) | up to the date of death (approximately 5 years)
The tolerance and the side effects of the treatment | every 3 weeks,up to completion of treatment(approximately 6 months)
  21 days(3 weeks) for one cycle,Toxicity was evaluated every cycle

OTHER OUTCOMES:
Epstein-Barr virus(EBV) DNA copies | every 3 weeks,up to completion of treatment(approximately 6 months)
  21 days(3 weeks) for one cycle
lymphocyte count | every 3 weeks,up to completion of treatment(approximately 6 months)
  21 days(3 weeks) for one cycle
Monocyte Count | every 3 weeks,up to completion of treatment(approximately 6 months)
  21 days(3 weeks) for one cycle
C reactive protein | every 3 weeks,up to completion of treatment(approximately 6 months)
  21 days(3 weeks) for one cycle
Plasma β2-microglobulin | every 3 weeks,up to completion of treatment(approximately 6 months)
  21 days(3 weeks) for one cycle
Urinary microglobulin β2 | every 3 weeks,up to completion of treatment(approximately 6 months)
  21 days(3 weeks) for one cycle

CONTACTS AND LOCATIONS:
Overall Officials: Wenqi Jiang, MD, Principal Investigator — Department of Medical Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, China State Key Laboratory of Oncology in South China, Sun Yat-Sen University Cancer Center, Guangzhou, China; Zhiming Li, MD, Principal Investigator — Department of Medical Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, China State Key Laboratory of Oncology in South China, Sun Yat-Sen University Cancer Center, Guangzhou, China
Locations (1):
- Department of Medical Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China